CLINICAL TRIAL: NCT03270644
Title: Effect of Lasmiditan on Heart Rate and Blood Pressure in Healthy Subjects Receiving Oral Doses of Propranolol
Brief Title: A Study of Lasmiditan and Propranolol in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 16857; H8H-MC-LAHD (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lasmiditan Reference (Experimental): Single oral dose of lasmiditan 200 mg on Day 1 as reference treatment.
  Interventions: Drug: Lasmiditan
- Propranolol Reference (Active Comparator): Twice-daily oral doses of propranolol 80 mg on Days 4-10 as reference treatment.
  Interventions: Drug: Propranolol
- Lasmiditan + Propranolol Test (Experimental): Single oral dose of lasmiditan 200 mg + two oral doses of propranolol 80 mg on Day 9 as test treatment.
  Interventions: Drug: Lasmiditan; Drug: Propranolol

INTERVENTIONS:
Drug: Lasmiditan — Administered orally
  Other Names: LY573144
  Arms: Lasmiditan + Propranolol Test; Lasmiditan Reference
Drug: Propranolol — Administered orally
  Arms: Lasmiditan + Propranolol Test; Propranolol Reference

SUMMARY:
This study will assess the effects on heart rate and blood pressure when a single dose of lasmiditan is administered with a daily dose of propranolol. This study will also measure how much lasmiditan gets into the bloodstream after taking lasmiditan alone and after taking it together with propranolol. The study will also look at how well both drugs are tolerated. Information about any side effects that may occur will be collected.

This study will last approximately 45 days including screening. This study will require 13 days/12 nights in a Clinical Research Unit (CRU) followed by 1 follow-up appointment approximately 7 days after the last dose. Screening is required within 28 days prior to the start of the study.

This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, as determined by medical history and physical examination
* Have a body mass index (BMI) of 19 to 35 kilograms per meter squared (kg/m²) inclusive, at the time of screening

Exclusion Criteria:

* Have known allergies to lasmiditan, propranolol, related compounds or any components of the formulation of lasmiditan or propranolol
* Have a history of, or electrocardiogram (ECG) findings of, clinically significant bradycardia, heart block, tachy or brady arrhythmias, sick sinus syndrome/sinoatrial block, or second or third-degree heart block, or have any other abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal supine blood pressure, defined as systolic blood pressure less than (<) 95 or greater than (>) 140 millimeters of mercury (mmHg) or diastolic blood pressure <65 or >90 mmHg at screening
* Have a supine pulse rate of <50 or >90 beats per minute (bpm) at screening
* Have an estimated glomerular filtration rate (eGFR) of <60 milliliter per minute (mL/min) per 1.73 meter squared (m2)
* Show evidence of significant active neuropsychiatric disease (for example, manic depressive illness, schizophrenia, depression)
* Show a history of central nervous system (CNS) conditions such as strokes, transient ischaemic attacks, significant head trauma, CNS infections, migraines, brain surgery or any other neurological conditions that, in the opinion of the investigator, increases the risk of participating in the study
* Are women with a positive pregnancy test or women who are lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Daytona Beach, Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Open-label fixed-sequence study in which participants received a single oral dose of lasmiditan 200 mg on Day (D) 1 Reference Treatment (R), then propranolol 80 mg administered orally twice daily from Day 4 through Day 10 Reference Treatment, with one single oral dose of lasmiditan 200 mg on Day 9 Test Treatment (T).
Groups:
- Lasmiditan (R); Propranolol (R) + Lasmiditan (T): Lasmiditan 200 mg single dose administered orally on D 1 (Reference); Propranolol 80 mg administered orally twice daily D4-10(Reference); Lasmiditan 200 mg administered orally on D9 (Test).
Period: Day 1 Lasmiditan Reference
Arm/Group | Lasmiditan (R); Propranolol (R) + Lasmiditan (T)
Started | 44
Received at Least One Dose of Study Drug | 44
Completed | 43
Not Completed | 1
Not completed — Physician Decision | 1
Period: Day 4 - 10 Propranolol Reference
Arm/Group | Lasmiditan (R); Propranolol (R) + Lasmiditan (T)
Started | 43
Received at Least One Dose of Study Drug | 43
Day 9 Lasmiditan + Propranolol Test | 42
Completed | 42
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Lasmiditan + Propranolol: Single 200 mg dose of lasmiditan administered orally on Day 1, then 80mg propranolol twice per day administered orally on Days 4 through 10, and 200 mg lasmiditan coadministered orally with propranolol on Day 9.
Arm/Group | Lasmiditan + Propranolol
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 28
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44
Mean Hourly Heart Rate [Mean (Standard Deviation); unit: beats per minute (BPM)] — Population: All participants who received one dose of study drug and had hourly HR baseline data.
  beats per minute (BPM)
    number analyzed (Participants) | 42
    (all) | 59.7 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day 8) in Mean Hourly Heart Rate Following Propranolol Administered Alone and When Coadministered With Lasmiditan
Description: Change from baseline in mean hourly heart rate recorded as beats per minute and collected by Holter ambulatory monitoring in response to propranolol administered alone and in combination with lasmiditan.
Time Frame: Baseline (Day 8), Day 9
Population: All participants who had at least one dose of study drug and had baseline and post-baseline cardiovascular measurements.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Groups:
- Propranolol (Reference Treatment): Propranolol 80 mg administered orally twice daily on Day 8.
- Lasmiditan + Propranolol (Test Treatment): Lasmiditan 200 mg coadministered with propranolol 80 mg on Day 9.
Arm/Group | Propranolol (Reference Treatment) | Lasmiditan + Propranolol (Test Treatment)
Number analyzed (Participants) | 42 | 42
beats per minute (bpm) | 59.7 (7.1) | 54.2 (5.8)
Statistical Analysis 1: Comparison: Propranolol (Reference Treatment) vs Lasmiditan + Propranolol (Test Treatment); Mean hourly HR was evaluated in a linear mixed-effects model with a fixed effect for treatment and a random effect for subject; Test type: Other; Difference of LSMeans = -5.45, 90% CI 2-sided [-7.27 to -3.64]

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Lasmiditan Alone and When Coadministered With Propranolol
Description: Maximum concentration of lasmiditan when administered alone on Day 1 and when coadministered with propranolol on Day 9.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose.
Population: All participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per mililiter (ng/mL)
Groups:
- Lasmiditan (Reference Treatment): Lasmiditan 200 mg single dose administered orally on Day 1.
- Lasmiditan + Propranolol (Test Treatment): Lasmiditan 200 mg coadministered orally with propranolol 80 mg on Day 9.
Arm/Group | Lasmiditan (Reference Treatment) | Lasmiditan + Propranolol (Test Treatment)
Number analyzed (Participants) | 44 | 42
nanogram per mililiter (ng/mL) | 323 (43) | 290 (31)
Statistical Analysis 1: Comparison: Lasmiditan (Reference Treatment) vs Lasmiditan + Propranolol (Test Treatment); Log-transformed PK parameters were evaluated in a linear mixed-effects model with a fixed effect for treatment and a random effect for subject; Test type: Other; Ratio of Geometric LSMeans = 0.884, 90% CI 2-sided [0.832 to 0.939]

3. Secondary Outcome: Pharmacokinetic: Maximum Observed Drug Concentration (Cmax) of Propranolol Alone and When Coadministered With Lasmiditan
Description: Maximum concentration of propranolol when administered alone on Day 8 and when coadministered with lasmiditan on Day 9.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose
Population: All participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Propranolol (Reference Treatment): Propranolol 80 mg administered orally twice daily Day 8.
- Lasmiditan + Propranolol (Test Treatment): Lasmiditan 200mg coadministered with 80 mg propranolol on Day 9.
Arm/Group | Propranolol (Reference Treatment) | Lasmiditan + Propranolol (Test Treatment)
Number analyzed (Participants) | 42 | 42
ng/mL | 133 (52) | 127 (43)
Statistical Analysis 1: Comparison: Propranolol (Reference Treatment) vs Lasmiditan + Propranolol (Test Treatment); Ratio of geometric LSMeans of Cmax used a mixed-effects repeated measures model adjusted for fixed effects for treatment, time point, time point by treatment, and random effect for subjects; Test type: Other; Ratio of Geometric LSMeans = 0.958, 90% CI 2-sided [0.917 to 1.00]

4. Secondary Outcome: Pharmacokinetic: Area Under the Concentration Versus Time Curve (AUC) From Time Zero to Last Measurable Concentration [AUC(0-tlast)] of Lasmiditan Alone and When Administered With Propranolol
Description: AUC versus time curve (AUC 0-tlast) of lasmiditan when administered alone on Day 1 and when coadministered with propranolol on Day 9.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose.
Population: All participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms * hour/mL (ng*h/mL)
Arm/Group | Lasmiditan (Reference Treatment) | Lasmiditan + Propranolol (Test Treatment)
Number analyzed (Participants) | 44 | 42
nanograms * hour/mL (ng*h/mL) | 2100 (39) | 2160 (30)
Statistical Analysis 1: Comparison: Lasmiditan (Reference Treatment) vs Lasmiditan + Propranolol (Test Treatment); [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio of Geometric LSMeans = 1.01, 90% CI 2-sided [0.967 to 1.04]

5. Secondary Outcome: Pharmacokinetic: Area Under the Concentration Versus Time Curve (AUC) of Propranolol During One Dosing Interval Alone and When Administered With Lasmiditan
Description: AUC versus time curve of propranolol during one dosing interval when administered alone on Day 8 and when administered with lasmiditan on Day 9.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose
Population: All participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Propranolol (Reference Treatment) | Lasmiditan + Propranolol (Test Treatment)
Number analyzed (Participants) | 42 | 42
ng*hr/mL | 910 (50) | 910 (43)
Statistical Analysis 1: Comparison: Propranolol (Reference Treatment) vs Lasmiditan + Propranolol (Test Treatment); [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio of Geometric LSMeans = 0.999, 90% CI 2-sided [0.967 to 1.03]

6. Secondary Outcome: Change From Baseline (Day 8) in PR Interval Following Propranolol Administered Alone and When Coadministered With Lasmiditan
Description: Change from baseline in PR interval, the interval between the P wave and the QRS complex calculated from electrocardiogram (ECG) data.
Time Frame: Baseline (Day 8), Day 9
Population: All participants who had at least one dose of study drug and had evaluable baseline and post-baseline cardiovascular measurements.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Propranolol (Reference Treatment) | Lasmiditan + Propranolol (Test Treatment)
Number analyzed (Participants) | 42 | 41
millisecond (msec) | 165.6 (20.5) | 161.9 (20.3)
Statistical Analysis 1: Comparison: Propranolol (Reference Treatment) vs Lasmiditan + Propranolol (Test Treatment); PR interval was evaluated in a linear mixed-effects model with a fixed effect for treatment and a random effect for subject; Test type: Other; Difference of LSMeans = -3.51, 90% CI 2-sided [-6.39 to -0.64]

7. Secondary Outcome: Change From Baseline (Day 8) in Systolic Blood Pressure Following Propranolol Administered Alone and When Coadministered With Lasmiditan
Description: Change from baseline in systolic blood pressure was measured in supine position.
Time Frame: Baseline (Day 8), Day 9
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Propranolol (Reference Treatment) | Lasmiditan + Propranolol (Test Treatment)
Number analyzed (Participants) | 42 | 42
millimeters of mercury (mmHg) | 106.9 (6.6) | 112.4 (10.9)
Statistical Analysis 1: Comparison: Propranolol (Reference Treatment) vs Lasmiditan + Propranolol (Test Treatment); Systolic blood pressure was evaluated in a linear mixed-effects model with a fixed effect for treatment and a random effect for subject; Test type: Other; Difference of LSMeans = 5.57, 90% CI 2-sided [3.57 to 7.57]

8. Secondary Outcome: Change From Baseline (Day 8) in Diastolic Blood Pressure Following Propranolol Administered Alone and When Coadministered With Lasmiditan
Description: Change from baseline in diastolic blood pressure was measured in supine position.
Time Frame: Baseline (Day 8), Day 9
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Propranolol (Reference Treatment) | Lasmiditan + Propranolol (Test Treatment)
Number analyzed (Participants) | 42 | 42
mmHg | 64.0 (6.2) | 67.4 (7.8)
Statistical Analysis 1: Comparison: Propranolol (Reference Treatment) vs Lasmiditan + Propranolol (Test Treatment); Diastolic blood pressure was evaluated in a linear mixed-effects model with a fixed effect for treatment and a random effect for subject; Test type: Other; Difference of LSMeans = 3.47, 90% CI 2-sided [1.99 to 4.95]

ADVERSE EVENTS:
Time Frame: Baseline through study completion (up to 23 days).
Description: All participants who have received at least one dose of study drug.
Groups:
- Lasmiditan 200 mg (Reference Treatment): Lasmiditan 200 mg single dose administered orally on Day 1.
- Propranolol 80 mg (Reference Treatment): Propranolol 80 mg administered orally twice daily on Day 4 to Day 10.
- Lasmiditan 200 mg + Propranolol 80 mg (Test Treatment): Lasmiditan 200 mg coadministered orally with propranolol 80 mg on Day 9.
Arm/Group | Lasmiditan 200 mg (Reference Treatment) | Propranolol 80 mg (Reference Treatment) | Lasmiditan 200 mg + Propranolol 80 mg (Test Treatment)
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/43 | 0/42
Other Adverse Events (participants affected / at risk) | 9/44 | 1/43 | 7/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lasmiditan 200 mg (Reference Treatment) (N=44) | Propranolol 80 mg (Reference Treatment) (N=43) | Lasmiditan 200 mg + Propranolol 80 mg (Test Treatment) (N=42)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lasmiditan 200 mg (Reference Treatment) (N=44) | Propranolol 80 mg (Reference Treatment) (N=43) | Lasmiditan 200 mg + Propranolol 80 mg (Test Treatment) (N=42)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 2 (2) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 6 (8) | 1 (1) | 4 (4)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT03270644/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03270644/SAP_001.pdf